CLINICAL TRIAL: NCT01257308
Title: Research of the EML4-ALK Gene Expression in the Pleural Effusion or Tumor Tissue From Lung Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Hsingjin Eugene Liu, MD PhD, Taipei Medical University WanFang Hospital
Other Study IDs: 99047
Record Dates: First submitted 2010-12-08; First posted 2010-12-09 (Estimated); Last update posted 2010-12-09 (Estimated); Status verified 2010-12

CONDITIONS: Lung Cancer Patients
Keywords: lung cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
We wants to analyse the EML4-ALK mutation rate in the patients who have non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* 20 or more than 20 years of age
* The pathological diagnosis confirmed lung cancer
* Patients have achieved pleural effusion, or surgical biopsy to obtain tumor tissue specimens
* The patient had signed inform consent

Exclusion Criteria:

* pleural effusion or tumor tissue can not be obtained
* the patient is not suitable to join the research according to the judgement by the investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung Cancer Patients
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-08; Study Completion 2013-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Hsin-Gjin Eugene Liu, Principal Investigator — Taipei Medical University WanFang Hospital
Locations (1):
- Taipei Medical University - WanFang Hospital, Taipei, Taiwan